CLINICAL TRIAL: NCT05413863
Title: A Randomised, Double-blind, Three-period, Partially Replicated Crossover, Euglycaemic Glucose Clamp Study in Healthy Volunteers to Demonstrate Pharmacokinetic and Pharmacodynamic Similarity of Biocon's Human Insulin R U-500 and Humulin® R U-500 (RHINE-4: Recombinant Human INsulin Equivalence-4)
Brief Title: Comparison of the Pharmacokinetic and Pharmacodynamic Properties of Biocon's Insulin R U-500 With Humulin® R U-500 (US Reference Product) in Healthy Subjects
Acronym: RHINE-4
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biocon Limited (Industry)
Collaborators: Profil Institut für Stoffwechselforschung GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: BIO-INS500-101
Record Dates: First submitted 2022-06-07; First posted 2022-06-10 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Healthy Volunteers
Keywords: Recombinant Human INsulin Equivalence-4; RHINE-4; Pharmacokinetic; Pharmacodynamic; Biocon's Insulin R U-500; Humulin® R U-500

STUDY DESIGN:
Intervention Model Description: Partially replicated design, crossover trial
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Sequence: Biocon's Human Insulin R U-500-Biocon's Human Insulin R U-500- Humulin® R U-500 (Experimental): Period 1:Biocon's Human Insulin R U-500 single subcutaneous dose of 0.3 IU/kg using a U-500 BD (Becton Dickinson) disposable syringe
  Period 2:Biocon's Human Insulin R U-500 single subcutaneous dose of 0.3 IU/kg using a U-500 BD (Becton Dickinson) disposable syringe
  Period 3:Humulin® R U-500 single subcutaneous dose of 0.3 IU/kg using a U-500 BD (Becton Dickinson) disposable syringe
  Interventions: Biological: Biocon's Human Insulin R U-500; Biological: Humulin® R U-500 (US Reference Product)
- Sequence: Biocon's Human Insulin R U-500-Humulin® R U-500- Humulin® R U-500 (Experimental): Period 1:Biocon's Human Insulin R U-500 single subcutaneous dose of 0.3 IU/kg using a U-500 BD (Becton Dickinson) disposable syringe
  Period 2:Humulin® R U-500 single subcutaneous dose of 0.3 IU/kg using a U-500 BD (Becton Dickinson) disposable syringe
  Period 3:Humulin® R U-500 single subcutaneous dose of 0.3 IU/kg using a U-500 BD (Becton Dickinson) disposable syringe
  Interventions: Biological: Biocon's Human Insulin R U-500; Biological: Humulin® R U-500 (US Reference Product)
- Sequence: Biocon's Human Insulin R U-500-Humulin® R U-500-Biocon's Human Insulin R U-500 (Experimental): Period 1:Biocon's Human Insulin R U-500 single subcutaneous dose of 0.3 IU/kg using a U-500 BD (Becton Dickinson) disposable syringe
  Period 2:Humulin® R U-500 single subcutaneous dose of 0.3 IU/kg using a U-500 BD (Becton Dickinson) disposable syringe
  Period 3:Biocon's Human Insulin R U-500 single subcutaneous dose of 0.3 IU/kg using a U-500 BD (Becton Dickinson) disposable syringe
  Interventions: Biological: Biocon's Human Insulin R U-500; Biological: Humulin® R U-500 (US Reference Product)
- Sequence: Humulin® R U-500-Biocon's Human Insulin R U-500-Biocon's Human Insulin R U-500 (Experimental): Period 1:Humulin® R U-500 single subcutaneous dose of 0.3 IU/kg using a U-500 BD (Becton Dickinson) disposable syringe
  Period 2:Biocon's Human Insulin R U-500 single subcutaneous dose of 0.3 IU/kg using a U-500 BD (Becton Dickinson) disposable syringe
  Period 3:Biocon's Human Insulin R U-500 single subcutaneous dose of 0.3 IU/kg using a U-500 BD (Becton Dickinson) disposable syringe
  Interventions: Biological: Biocon's Human Insulin R U-500; Biological: Humulin® R U-500 (US Reference Product)
- Sequence: Humulin® R U-500 -Biocon's Human Insulin R U-500-Humulin® R U-500 (Experimental): Period 1:Humulin® R U-500 single subcutaneous dose of 0.3 IU/kg using a U-500 BD (Becton Dickinson) disposable syringe
  Period 2:Biocon's Human Insulin R U-500 single subcutaneous dose of 0.3 IU/kg using a U-500 BD (Becton Dickinson) disposable syringe
  Period 3:Humulin® R U-500 single subcutaneous dose of 0.3 IU/kg using a U-500 BD (Becton Dickinson) disposable syringe
  Interventions: Biological: Biocon's Human Insulin R U-500; Biological: Humulin® R U-500 (US Reference Product)
- Sequence: Humulin® R U-500-Humulin® R U-500-Biocon's Human Insulin R U-500 (Experimental): Period 1:Humulin® R U-500 single subcutaneous dose of 0.3 IU/kg using a U-500 BD (Becton Dickinson) disposable syringe
  Period 2:Humulin® R U-500 single subcutaneous dose of 0.3 IU/kg using a U-500 BD(Becton Dickinson) disposable syringe
  Period 3:Biocon's Human Insulin R U-500 single subcutaneous dose of 0.3 IU/kg using a U-500 BD (Becton Dickinson) disposable syringe
  Interventions: Biological: Biocon's Human Insulin R U-500; Biological: Humulin® R U-500 (US Reference Product)

INTERVENTIONS:
Biological: Biocon's Human Insulin R U-500 — Biocon's Human Insulin R U-500 (Insulin Human Injection 500 units/mL), 3 mL cartridges (containing 1,500 units of insulin).
Biological: Humulin® R U-500 (US Reference Product) — Humulin® R U-500 (US Reference Product), 3 mL single-patient-use KwikPen® (containing 1,500 units of insulin)

SUMMARY:
Single-centre, randomised, double-blind, three-period, six-sequence, partially replicated design, crossover trial in healthy subjects

DETAILED DESCRIPTION:
The present study is designed to demonstrate pharmacokinetic and pharmacodynamic equivalence of Biocon's Human Insulin R U-500 with Humulin® R U-500 in healthy subjects.

The treatment consists of one single dose of the test or reference product, administered during each of the three study periods, separated by 5-7 days between each dosing. The planned trial duration for each subject is about 18 to 44 days. Eligible subjects will undergo three euglycaemic clamp examinations (each of 24 hours duration).

Depending on the sequence in which a particular subject is randomized, each subject will either undergo two clamps with administration of test product plus one clamp with administration of reference product, or, two clamps with administration of reference product plus one clamp with administration of test product, in random order.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or post-menopausal female subjects. The post-menopausal state is defined as no menses for 12 months without an alternative medical cause and confirmed by a follicle stimulating hormone (FSH) level in the post-menopausal range (≥ 25.8 IU/L).
* Age between 18 and 55 years, both inclusive.
* Body Mass Index (BMI) between 18.5 and 29.0 kg/m2, both inclusive.
* Fasting plasma glucose concentration ≤ 100 mg/dL.
* Considered generally healthy upon completing the medical history and screening safety assessments, as judged by the Investigator.

Exclusion Criteria:

* Known or suspected hypersensitivity to investigational medicinal products (IMPs) or related products.
* Receipt of any medicinal product in clinical development within 30 days or five times its half-life (whichever is longer) before randomisation in this trial.
* Systolic blood pressure < 90 mmHg or > 139 mmHg and/or diastolic blood pressure < 50 mmHg or > 89 mmHg after resting for at least 5 minutes in the supine position (excluding white-coat hypertension; therefore, a repeat test showing results within range will be acceptable).
* Pulse rate at rest outside the range of 50-90 beats per minute.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2022-05-30 (Actual); Primary Completion 2022-12-12 (Actual); Study Completion 2022-12-12 (Actual)

PRIMARY OUTCOMES:
Primary pharmacokinetics (PK) endpoint: area under the insulin concentration curve(AUCins).0-12h | 0 to12 hours
  Area under the insulin concentration curve
Primary pharmacokinetics (PK) endpoint: maximum observed insulin concentration(Cins.max) | NAP (Not Applicable)
  Maximum observed insulin concentration
Primary pharmacodynamics (PD) endpoint:area under the glucose infusion rate curve (AUCGIR)0-12h | 0 to 12 hours
  Area under the glucose infusion rate curve
Primary pharmacodynamics (PD) endpoint:maximum observed glucose infusion rate (GIRmax) | NAP (Not Applicable)
  Maximum observed glucose infusion rate

SECONDARY OUTCOMES:
Secondary pharmacokinetics (PK) endpoint: area under the insulin concentration-time curve(AUCins).0-infinity | 0 hours to 24 hours
  Area under the insulin concentration-time curve
Secondary pharmacokinetics (PK) endpoint: area under the insulin concentration-time curve(AUCins).0-24h | 0 to 24 hours
  Area under the insulin concentration-time curve
Secondary pharmacokinetics (PK) endpoint: area under the insulin concentration-time curve (AUCins).12-24h | 12 to 24 hours
  Area under the insulin concentration-time curve
Secondary pharmacokinetics (PK) endpoint:time to maximum observed insulin concentration (tmax.ins) | 0 to 24 hours
  Time to maximum observed insulin concentration
Secondary pharmacokinetics (PK) endpoint:terminal elimination rate constant of insulin (λz) | 0 to 24 hours
  Terminal elimination rate constant of insulin
Secondary pharmacokinetics (PK) endpoint: terminal elimination half-life (t½) | 0 to 24 hours
  Terminal elimination half-life calculated
Secondary pharmacokinetics (PK) endpoint: time(t)50%-Insulin (INS)(early) | 0 to 24 hours
  Time to half-maximum before Cmax
Secondary pharmacokinetics (PK) endpoint: time(t) 50%-Insulin (INS)(late) | 0 to 24 hours
  Time to half-maximum after Cmax
Secondary pharmacodynamics (PD) endpoint: areas under the glucose infusion rate curve(AUCGIR).0-24h | 0 to 24 hours
  Area under the glucose infusion rate curve
Secondary pharmacodynamics (PD) endpoint: areas under the glucose infusion rate curve(AUCGIR).12-24h | 12 to 24 hours
  Area under the glucose infusion rate curve
Secondary pharmacodynamics (PD) endpoint: time to maximum glucose infusion rate(tmax.GIR) | 0 to 24 hours
  Time to maximum glucose infusion rate
Secondary pharmacodynamics (PD) endpoint:time to half-maximum glucose infusion rate before GIRmax (tGIR.50%-early) | 0 to 24 hours
  Time to half-maximum glucose infusion rate before GIRmax
Secondary pharmacodynamics (PD) endpoint: time to half-maximum glucose infusion rate after GIRmax (tGIR.50%-late) | 0 to 24 hours
  Time to half-maximum glucose infusion rate after GIRmax
Secondary pharmacodynamics (PD) endpoint: Onset of action, time from trial product administration until plasma glucose concentration has decreased at least 5 mg/dL from baseline, | 0 to 24 hours
  Time from trial product administration until plasma glucose concentration

OTHER OUTCOMES:
Safety endpoint: Number of subjects with Adverse Events (AEs) | Signing of Informed consent form (ICF) to follow-up period (Total duration: 44 days approximate)
Safety endpoint: Number of subjects with Clinically significant changes in Physical examination | Signing of Informed consent form (ICF) to follow-up period (Total duration: 44 days approximate)
Safety endpoint: Number of subjects with Clinically significant changes in Vital signs | Signing of Informed consent form (ICF) to follow-up period (Total duration: 44 days approximate)
Safety endpoint: Local tolerability assessment / Injection site reactions | Signing of Informed consent form (ICF) to follow-up period (Total duration:44 days approximate)
  Number of subjects with Injection Site Reactions
Safety endpoint: Number of subjects with clinically significant changes in Laboratory safety parameters | Signing of Informed consent form (ICF) to follow-up period (Total duration:44 days approximate)
Safety endpoint: Number of subjects with clinically significant changes in ECG | Signing of Informed consent form (ICF) to follow-up period (Total duration:44 days approximate)

CONTACTS AND LOCATIONS:
Overall Officials: Dr Ulrike Hövelmann, MD, Principal Investigator — Profil Institut für Stoffwechselforschung GmbH
Locations (1):
- Profil Institut für Stoffwechselforschung GmbH 9, Neuss, Germany

IPD SHARING:
Plan to Share IPD: No